CLINICAL TRIAL: NCT01964066
Title: Effectiveness of Thoracic Epidural Analgesia for the Prevention of Post-ERCP Pancreatitis
Brief Title: Study of Effectiveness of Thoracic Epidural Analgesia for the Prevention of Acute Pancreatitis After ERCP Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Volgograd State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 124/2007/12/24
Record Dates: First submitted 2013-09-17; First posted 2013-10-17 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2013-10

CONDITIONS: Post-ERCP Acute Pancreatitis
Keywords: therapeutic ERCP; prevention of post-ERCP pancreatitis; thoracic epidural analgesia
MeSH Terms: interventions — Cholangiopancreatography, Endoscopic Retrograde; Tea; Analgesia, Epidural; Anesthesia, Epidural; Premedication; Balanced Anesthesia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ERCP & Thoracic epidural analgesia (Experimental): Used thoracic epidural analgesia (ropivacaine 0.5% -10ml) for pain relief ERCP.
  Interventions: Procedure: ERCP; Procedure: Thoracic epidural analgesia
- ERCP & Premedication (Active Comparator): Used Premedication (trimeperidine 2% -1ml intravenously) for pain control ERCP.
  Interventions: Procedure: ERCP; Procedure: Premedication

INTERVENTIONS:
Procedure: ERCP — Endoscopic retrograde cholangiopancreatography balloon dilatation
  Other Names: endoscopic transpapillary intervention
Procedure: Thoracic epidural analgesia — Thoracic epidural analgesia between thoracic vertebrae VII-VIII (Ropivacaine 0.5%-10ml)
  Other Names: Epidural analgesia; Epidural anaesthesia
  Arms: ERCP & Thoracic epidural analgesia
Procedure: Premedication — For premedication used trimeperidine 2%-1ml intravenously.
  Other Names: anociassociation; anocithesia; prenarcosis
  Arms: ERCP & Premedication

SUMMARY:
For 40 years, the post-ERCP (endoscopic retrograde cholangiopancreatography) pancreatitis has been the most frequent adverse effect of endoscopic transpapillary interventions. We sought to determine the efficacy of thoracic epidural analgesia for the prevention of post-ERCP pancreatitis.

Between 2008 and 2013, a randomized study of the results of endoscopic treatment of 491 patients was conducted. The first group of patients (N=247) received thoracic epidural analgesia (TEA) during ERCP procedures, the patients of the second group (N=244) received a narcotic analgesic. To detect statistically significant differences between research groups adjusted odds ratios (OR) and their 95% confidence interval (CI) were calculated.

DETAILED DESCRIPTION:
Preoperatively the subjects were randomly assigned (by using sealed envelopes - blind randomization) into two groups, 250 patients each.

The patients of the first group had TEA applied during the ERCP procedure; other methods of pain relief were applied to the patients of the second (control) group.

The first group (TEA group) of patients received the following premedication: atropine sulfate 0.5-1 mg, midazolan 5 mg. The puncture and catheterization of the epidural space was carried out according to standard procedure between thoracic vertebrae VII-VIII. Half an hour before performing ERCP ropivacaine 0.5% -10 ml. was injected into the epidural space.

The second group (control group) of patients received the following premedication: atropine sulfate 0.5 -1 mg, midazolan 5 mg, trimeperidine 2% -1 ml.

ELIGIBILITY:
Inclusion criteria:

* Patients with performed therapeutic ERCP;
* The ERCP procedure was performed in a patient for the first time;
* Prior to the ERCP procedure the patient didn't have any clinical signs of acute pancreatitis.

Exclusion criteria:

- Development of complications during the ERCP procedure that required urgent surgical intervention (massive haemorrhage, Dormia basket avulsion and others).

Ages: 15 Years to 92 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 491 (Actual)
Dates: Start 2008-01; Primary Completion 2013-03 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
the prevention of post-ERCP pancreatitis | one day

CONTACTS AND LOCATIONS:
Overall Officials: Mihail Turovets, PhD, Study Chair — Clinic №1 of Volgograd state medical university
Locations (1):
- Clinic №1 of Volgograd State Medical University, Volgograd, Russia